CLINICAL TRIAL: NCT06082388
Title: Comparison of the Clinical Utility of Atropine and Isoprenaline in the Invasive Diagnosis of Arrhythmias
Brief Title: Atropine vs Isoprenaline in the Invasive Diagnosis of Arrhythmias
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Medical University of Lodz (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: RNN/327/20/KE
Record Dates: First submitted 2022-01-12; First posted 2023-10-13 (Actual); Last update posted 2023-10-13 (Actual); Status verified 2023-10

CONDITIONS: Cardiac Arrhythmia; Supraventricular Arrhythmia
Keywords: Electrophysiological study; Atropine; Isoprenaline; Supraventricular arrhythmia; Ablation
MeSH Terms: conditions — Arrhythmias, Cardiac | interventions — Isoproterenol

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Atropine (Active Comparator): Patients in whom during electrophysiological study atropine will be used. I.v. bolus of 0.01 mg/kg b.w. will be administered to reach the increase of heart rate of 25% or up to 130/min. If necessary, dose will be increased every 5 minutes until mention above parameters are achieved. Maximum dose will be 0.4 mg/kg b.w.
  Interventions: Drug: Comparison of atropine and isoprenaline
- Isoprenaline (Active Comparator): Patients in whom during electrophysiological study isoprenaline will be used. Continuous i.v. infusion of 0.01 mcg/kg b.w./min will be administered to reach the increase of heart rate of 25% or up to 130/min. If necessary, dose will be doubled every 5 minutes until mention above parameters are achieved. Maximum dose will be 20 mcg/min.
  Interventions: Drug: Comparison of atropine and isoprenaline

INTERVENTIONS:
Drug: Comparison of atropine and isoprenaline — Comparison of heart conductive system and arrhythmia inducibility after using atropine or isoprenaline

SUMMARY:
During electrophysiological study (EPS) multiple drugs are used to reveal arrhythmias and/or conductive system disorders. Two most often used agents are atropine and isoprenaline. Due to their distinct pharmacological properties, they are affecting myocardium in different manner. Those dissimilarities can affect the EPS course and long-term prognosis. The aim of presented study is to evaluate the optimal protocol of pharmacotherapy during EPS.

DETAILED DESCRIPTION:
Electrophysiological study (EPS) is essential tool for heart rhythm disorders diagnostic. Inducibility of arrhythmia before ablation to confirm the diagnosis and inability to do so after the procedure is crucial for long-term success. Multiple drugs are used to reveal arrhythmias and/or conductive system disorders. Two most often used are atropine and isoprenaline. Atropine is a natural, selective antagonist of cholinergic receptors M1 and M2. It reverses the inhibitory effect of vagal nerve on myocardium. This improves sinus node automatism and conduction in atrioventricular node. Isoprenaline is a preferential agonist of beta-1-adrenergic receptors. It has bathmotropic and chronotropic effect. During daily clinical practice those two drugs are often used interchangeably. However, differences in pharmacokinetics and pharmacodynamics may affect the results. There are lack of data directly comparing those two agents. There are isolated evidences that arrhythmia inducibility rate after the ablation differs between those two drugs. This may lead to the misconception of ablation as successful. The aim of presented study is to evaluate the optimal protocol of pharmacotherapy during EPS.

ELIGIBILITY:
Inclusion Criteria:

* Patients with indication for electrophysiological study according to present guidelines of European Society of Cardiology

Exclusion Criteria:

* Not willing or incapable to give written informed consent.
* Previous diagnosed ventricle tachycardia or fibrillation
* Previous diagnosed atrial fibrillation or flutter
* Glaucoma (contraindication for atropine)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2023-11-09 (Estimated); Primary Completion 2025-09 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Evaluation of sino-atrial conduction time | During the procedure
  Sino-atrial conduction time (ms) during programed atrial stimulation will be assessed to examine the function of sinus node.
Evaluation of sinus node recovery time | During the procedure
  Sinus node recovery time (ms) during programed atrial stimulation will be assessed to examine the function of sinus node.
Evaluation of anterograde atrioventricular conduction | During the procedure
  Anterograde Wenkebach point (ms) and effective refractory period of atrioventricular node (ms) during programed atrial stimulation will be assessed.
Evaluation of retrograde atrioventricular conduction | During the procedure
  Retrograde Wenkebach point (ms) and effective refractory period of atrioventricular node (ms) during programed ventricular stimulation will be assessed.
Arrhythmia inducibility | During the procedure
  Inducibility of anticipated arrythmia before and after drug administration and after eventual ablation.
Long-term success rate | 12 months
  Recurrence of clinical arrhythmia during 12 months of observation

SECONDARY OUTCOMES:
Incidence of adverse events during the electrophysiological study. | During the procedure
  Analysis of adverse events during the electrophysiological study according to used drug. Adverse events includes: death, stroke, cardiogenic shock, anaphylaxis, myocardial infarction, electric storm.
Incidence of adverse events during the 12-month follow up. | 12 months
  Analysis of adverse events during the 12-month follow up according to used drug. Adverse events includes: death, stroke, cardiogenic shock, anaphylaxis, myocardial infarction, electric storm.
Length of the procedure | During the procedure
  Analysis of the whole procedure time according to used drug.
Procedure time form drug administration till the end. | During the procedure
  Analysis of the procedure time form atropine/isoprenaline administration till the end.

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Electrocardiology Medical University of Lodz, Lodz, Poland

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Result] Stellbrink C, Diem B, Schauerte P, Brehmer K, Schuett H, Hanrath P. Differential effects of atropine and isoproterenol on inducibility of atrioventricular nodal reentrant tachycardia. J Interv Card Electrophysiol. 2001 Dec;5(4):463-9. doi: 10.1023/a:1013258331023. PMID 11752915
- [Result] Toda I, Kawahara T, Murakawa Y, Nozaki A, Kawakubo K, Inoue H, Sugimoto T. Electrophysiological study of young patients with exercise related paroxysms of palpitation: role of atropine and isoprenaline for initiation of supraventricular tachycardia. Br Heart J. 1989 Mar;61(3):268-73. doi: 10.1136/hrt.61.3.268. PMID 2930664
- [Result] Hatzinikolaou H, Rodriguez LM, Smeets JL, Timmermans C, Vrouchos G, Grecas G, Wellens HJ. Isoprenaline and inducibility of atrioventricular nodal re-entrant tachycardia. Heart. 1998 Feb;79(2):165-8. doi: 10.1136/hrt.79.2.165. PMID 9538310